CLINICAL TRIAL: NCT04489121
Title: The Efficacy of Preseasonal Omalizumab Treatment in Seasonal Allergic Rhinitis Patients
Brief Title: The Efficacy of Preseasonal Omalizumab Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Luo Zhang, President, Beijing TongRen Hospital, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Preseasonal-OMA-AR
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Omalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omalizumab preseasonal treatment (Experimental): For patients in the Omalizumab group, subcutaneous injections of Omalizumab based on the specific participant's weight and serum total IgE was performed 2 weeks prior the anticipated pollen season. Rescue medication could be used during pollen seasons.
  Interventions: Drug: Omalizumab
- control (No Intervention): No preseasonal treatment was performed. Rescue medication could be used during pollen seasons.

INTERVENTIONS:
Drug: Omalizumab — For patients in the Omalizumab group, subcutaneous injections of Omalizumab based on the specific participant's weight and serum total IgE was performed 2 weeks prior the anticipated pollen season.
  Arms: omalizumab preseasonal treatment

SUMMARY:
Allergic rhinitis (AR) is induced by an immunoglobulin E (IgE)-mediated reaction in the allergen-sensitized subjects, affecting 10% to 40% of the world population. AR could be divided into two kinds, perennial AR and seasonal AR (SAR).

In recent years, biologics have become promising drugs for allergic diseases. The efficacy and safety of Omalizumab in treating SAR have been well proven by previous studies. However, the efficacy in preseasonal treatment for SAR has not yet been studied before.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 to 60 years (inclusive).
* With history of SAR for at least two years, with/without conjunctivitis and without asthma
* Two or more nasal symptoms scores were ≥ 2 points during July - October in the last year.
* Sensitised to common autumn pollens including sagewort and ragweed (a specific IgE level ≥ 3.5 kU/L).
* Patients who have been informed of the nature and aims of the study and have given their written consent, willing to comply with the protocol.
* Patients who are able to understand the information given and the consent and complete the daily record card.

Exclusion Criteria:

* Patients with oral diseases/ allergies within the run-in period.
* Patients accepted any kind of operations within 4 weeks of the run-in period.
* Patients applied for systemic glucocorticoids within 4 weeks in the run-in period.
* Patients with PAR.
* Patients with any nasal condition that could confound the results of the study (chronic rhinitis, chronic rhinosinusitis with/without polyps).
* Whatever the co-sensitization leading to clinically relevant AR, conjunctivitis or asthma likely to significantly change the symptoms of the patient throughout the study.
* patients with comorbidity of severe asthma.
* Patients applying beta-antagonist (local or systemic appliance).
* Pregnant, breast-feeding / sexually active women of childbearing potential.
* Patients treated with AIT for pollens within 3 years.
* Participation in any clinical study within the 3 months of the run-in period.
* Patients at risk of non-compliance..
* Patients with immunologic suppression, diabetes mellitus, autonomic neuropathy, coronary heart disease or hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
the change of total nasal symptoms scores | at baseline, week 2 (the initial phase of pollen season) , week 4(during the anticipated peak pollen phase), and week 6 (the end of season).
Rescue medication score | at week 2 (the initial phase of pollen season) , week 4(during the anticipated peak pollen phase), and week 6 (the end of season).
  when the symptoms were very severe and could not tolerated, the patients could use loratadine as rescue medication.
  The need for rescue medication was assessed as rescue medication score (RMS), analyzed as the weekly sum of daily use of Loratadine (10mg/d, equivalent to 1 point) or nasal corticosteroid spray (2 points)

SECONDARY OUTCOMES:
the change of quality of life | at baseline, week 2 (the initial phase of pollen season) , week 4(during the anticipated peak pollen phase), and week 6 (the end of season).
  mini Rhinoconjunctivitis Quality of Life Questionnaire (miniRQLQ)
adverse events | one hour after injection in the Omalizumab group
  Any adverse event following injection was assessed by physicians and patients. Patients in the Omalizumab group are instructed to record any unexpected signs, symptoms, and feelings during the subcutaneous injection of Omalizumab.
eosinophilic indicators in nasal secretions | at baseline, week 2 (the initial phase of pollen season) , week 4(during the anticipated peak pollen phase), and week 6 (the end of season).
  The level of eosinophilic indicators; Charcot-Leyden crystal (CLC) , Cystatin SN

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China